CLINICAL TRIAL: NCT01761240
Title: A Phase I Study of the Safety, Tolerability, and Pharmacokinetics of MORAb-066, a Humanized Monoclonal Antibody to Human Tissue Factor, in Patients With Advanced or Metastatic Breast, Pancreatic, Colorectal, or Non-Small Cell Lung Cancer (Adenocarcinoma) Malignancies
Brief Title: Dose Escalation Study MORAb-066 Targeting Tissue Factor (TF)-Expressing Malignancies Including Breast, Pancreatic, Colorectal, NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Morphotek (Industry)
Collaborators: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MORAb-066-001
Record Dates: First submitted 2013-01-03; First posted 2013-01-04 (Estimated); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer; Pancreatic Cancer; Colorectal Cancer; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- MORAb-066 0.1 mg/kg (Experimental): Participants will receive MORAb-066 0.1 milligram per kilogram (mg/kg), infusion intravenously, on Days 1, 8, 15, and 22, in each 28-day treatment cycle until disease progression, participant's discontinuation due to unacceptable toxicity, withdrawal by participants, or discontinuation by study physician decision.
  Interventions: Drug: MORAb-066
- MORAb-066 0.3 mg/kg (Experimental): Participants will receive MORAb-066 0.3 mg/kg, infusion intravenously, on Days 1, 8, 15, and 22, in each 28-day treatment cycle until disease progression, the participant discontinuation due to unacceptable toxicity, withdrawal by participants, or discontinuation by study physician decision.
  Interventions: Drug: MORAb-066
- MORAb-066 1 mg/kg (Experimental): Participants will receive MORAb-066 1 mg/kg, infusion intravenously, on Days 1, 8, 15, and 22, in each 28-day treatment cycle until disease progression, the participant's discontinuation due to unacceptable toxicity, withdrawal by participants, or discontinuation by study physician decision.
  Interventions: Drug: MORAb-066
- MORAb-066 2 mg/kg (Experimental): Participants will receive MORAb-066 2 mg/kg, infusion intravenously, on Days 1, 8, 15, and 22, in each 28-day treatment cycle until disease progression, the participant's discontinuation due to unacceptable toxicity, withdrawal by participants, or discontinuation by study physician decision.
  Interventions: Drug: MORAb-066
- MORAb-066 3 mg/kg (Experimental): Participants will receive MORAb-066 3 mg/kg, infusion intravenously, on Days 1, 8, 15, and 22, in each 28-day treatment cycle until disease progression, the participant discontinuation due to unacceptable toxicity, withdrawal by participants, or discontinuation by study physician decision.
  Interventions: Drug: MORAb-066

INTERVENTIONS:
Drug: MORAb-066 — MORAb-066 infusion.

SUMMARY:
This study is a Phase I, first in human, dose-escalation study of MORAb-066, an investigational humanized immunoglobulin G (IgG) monoclonal antibody (mAb) that targets TF-expressing malignancies that include breast, pancreatic, colorectal, and non-small-cell lung cancer (NSCLC) (adenocarcinoma). This open-label study will assess the safety, tolerability, and pharmacokinetics of MORAb-066 administered weekly. This study will identify the maximum tolerated dose (MTD) when MORAb-066 is administered IV once weekly on a 28-day cycle.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria in order to be included in this clinical trial:

1. Histologically or cytologically confirmed diagnosis of breast, colorectal, pancreas, or NSCLC (adenocarcinoma) that is metastatic or unresectable for which there is no effective therapy.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1 (see Appendix A).
3. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
4. Subject has recovered (to Grade less than or equal to 1) from all clinically significant toxicities related to prior antineoplastic therapies with the exception of alopecia and bone marrow and organ functions (described separately below).
5. Adequate organ system function less than or equal to 2 weeks prior to Day1, defined as follows:

   * Absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/L
   * Platelets greater than or equal to 100 x 10^9/L
   * Hemoglobin greater than or equal to 9 g/dL
   * Prothrombin time/partial thromboplastin time (PT/PTT) within institutional limits of normal
   * Serum total bilirubin less than or equal to 1.5 times the upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 3.0 x ULN if no liver involvement or less than or equal to 5 x ULN with liver involvement.
   * Serum creatinine less than or equal to 1.5 x ULN or calculated creatinine clearance greater than or equal to 50 mL/min as calculated by the Cockcroft-Gault method, OR 24-hour measured urine creatinine clearance greater than or equal to 50 mL/min.
6. Life expectancy of greater than or equal to 12 weeks.
7. Female patients of child-bearing potential (see Appendix C), and all male patients must consent to use a medically acceptable method of contraception throughout the study period and for 30 days after their last MORAb-066 administration. A barrier method of contraception must be included.
8. Patients must be greater than or equal to 18 years of age.
9. Patients entering this study will be asked to provide archival tissue from a previous tumor biopsy (if available) for correlative testing. If tissue is not available, the subject will still be eligible for enrollment into the study.
10. Ability to understand the nature of this study and give written informed consent.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from trial entry:

1. Patients currently receiving cancer therapy (i.e., chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, surgery and/or tumor embolization).
2. Use of an investigational drug within 21 days or 5 half-lives (whichever is shorter) prior to the first dose of MORAb-066. For investigational drugs for which 5 half-lives is less than 21 days, a minimum of 10 days between termination of the investigational drug and administration of MORAb-066 is required.
3. Any major surgery, chemotherapy, radiotherapy, or immunotherapy within the last 21 days (limited palliative radiation is allowed greater than or equal to 2 weeks).
4. Subject has received wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) less than or equal to 28 days or limited field radiation for palliation less than or equal to 14 days prior to starting study drug or has not recovered from side effects of such therapy.
5. Known intracranial involvement, leptomeningeal metastases or spinal cord compression due to disease.
6. Known allergy or hypersensitivity to monoclonal antibodies.
7. Known bleeding diathesis, such as factor deficiency, factor inhibitor, platelet disorder, or who are on active anticoagulation, or any dose of aspirin within 5 days prior to first dose of MORAb-066.
8. Known prior significant bleeding history.
9. Patients with ureteral stents or 3+ blood in the urine at baseline.
10. Patients who are receiving chronic systemic anticoagulation therapy (warfarin sodium or heparin, etc.).
11. Patients who received a previous mAb therapy and have evidence of an immune or allergic reaction or previously documented HAHA reaction.
12. A serious non-healing wound, active ulcer, or untreated bone fracture. An abdominal fistula or gastrointestinal perforation less than 6 months prior to treatment.
13. History of hematemesis or hemoptysis (defined as having bright red blood of 1/2 teaspoon or more per episode) less than or equal to 1 month prior to study enrollment.
14. Subject has cardiac dysfunction including any of the following:

    * Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular ejection fraction function
    * QTcF greater than 470 msec
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV [see Appendix B])
    * Angina not well-controlled by medication
15. A serious active infection (bacterial or fungal) at the time of treatment, or another serious underlying medical condition that would impair the ability of the subject to receive protocol treatment.
16. Chronic inflammatory disorder(e.g., inflammatory bowel disease, active vasculitis).
17. Herbal preparations/medications must be discontinued 7 days prior to first dose of study drug (see Section 5.3.1).
18. Known diagnosis of human immunodeficiency virus, Hepatitis B or Hepatitis C.
19. History or current diagnosis of glomerulonephritis
20. History of clinically significant or current diagnosis of hematuria.
21. Women who are pregnant or lactating.
22. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
23. Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol.
24. Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-06-19 (Actual); Primary Completion 2016-02-09 (Actual); Study Completion 2016-02-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 19 June 2013 to 09 February 2016.
Pre-assignment Details: A total of 27 participants were enrolled and treated in the study.
Groups:
- MORAb-066 0.1 mg/kg: Participants received MORAb-066 0.1 milligram per kilogram (mg/kg), infusion intravenously, on Days 1, 8, 15, and 22, in each 28-day treatment cycle until disease progression, participant's discontinuation due to unacceptable toxicity, withdrawal by participants, or discontinuation by study physician decision.
- MORAb-066 0.3 mg/kg: Participants received MORAb-066 0.3 mg/kg, infusion intravenously, on Days 1, 8, 15, and 22, in each 28-day treatment cycle until disease progression, the participant discontinuation due to unacceptable toxicity, withdrawal by participants, or discontinuation by study physician decision.
- MORAb-066 1 mg/kg: Participants received MORAb-066 1 mg/kg, infusion intravenously, on Days 1, 8, 15, and 22, in each 28-day treatment cycle until disease progression, the participant's discontinuation due to unacceptable toxicity, withdrawal by participants, or discontinuation by study physician decision.
- MORAb-066 2 mg/kg: Participants received MORAb-066 2 mg/kg, infusion intravenously, on Days 1, 8, 15, and 22, in each 28-day treatment cycle until disease progression, the participant's discontinuation due to unacceptable toxicity, withdrawal by participants, or discontinuation by study physician decision.
- MORAb-066 3 mg/kg: Participants received MORAb-066 3 mg/kg, infusion intravenously, on Days 1, 8, 15, and 22, in each 28-day treatment cycle until disease progression, the participant discontinuation due to unacceptable toxicity, withdrawal by participants, or discontinuation by study physician decision.
Period: Overall Study
Arm/Group | MORAb-066 0.1 mg/kg | MORAb-066 0.3 mg/kg | MORAb-066 1 mg/kg | MORAb-066 2 mg/kg | MORAb-066 3 mg/kg
Started | 3 | 4 | 5 | 7 | 8
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 5 | 7 | 8
Not completed — Progressive disease:radiology assessment | 3 | 3 | 0 | 0 | 0
Not completed — Progressive disease:clinical assessment | 0 | 0 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 6
Not completed — Death | 0 | 1 | 1 | 2 | 1
Not completed — Non-compliance | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who had received at least 1 dose of study drug.
Groups:
- MORAb-066 0.1 mg/kg: Participants received MORAb-066 0.1 mg/kg, infusion intravenously, on Days 1, 8, 15, and 22, in each 28-day treatment cycle until disease progression, participant's discontinuation due to unacceptable toxicity, withdrawal by participants, or discontinuation by study physician decision.
- Total: Total of all reporting groups
Arm/Group | MORAb-066 0.1 mg/kg | MORAb-066 0.3 mg/kg | MORAb-066 1 mg/kg | MORAb-066 2 mg/kg | MORAb-066 3 mg/kg | Total
Number analyzed (Participants) | 3 | 4 | 5 | 7 | 8 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (7.21) | 57.8 (9.39) | 55.2 (6.06) | 62.4 (7.98) | 64.3 (8.75) | 60.8 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 4 | 4 | 15
  Male | 1 | 2 | 2 | 3 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 5 | 6 | 7 | 24
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 1 | 0 | 3
  White | 3 | 4 | 2 | 5 | 8 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Safety assessments consisted of monitoring and recording all AEs and SAEs; regular monitoring of hematology, blood chemistry, urine values, and vital signs; periodic measurement of electrocardiograms (ECGs) and Eastern Cooperative Oncology Group (ECOG) assessments; and performance of physical examinations.
Time Frame: First dose of study drug (Baseline) up to 30 days after last dose of study drug (Up to approximately 2 years 7 months)
Population: The safety analysis set was the group of participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-066 0.1 mg/kg | MORAb-066 0.3 mg/kg | MORAb-066 1 mg/kg | MORAb-066 2 mg/kg | MORAb-066 3 mg/kg
Number analyzed (Participants) | 3 | 4 | 5 | 7 | 8
Participants
  TEAEs | 3 | 4 | 5 | 7 | 8
  SAEs | 0 | 1 | 3 | 4 | 3

2. Secondary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: DLT was defined using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 as any grade 3 or 4 hematemesis, hemoptysis, hematochezia, bright red blood per rectum, epistaxis, gingival bleeding, hemarthrosis, haematuria, uncontrollable menses, or any other bleeding thought to be significant as per assessment of the investigator, regardless of grade.
Time Frame: Cycle 1 (Cycle length=28 days)
Population: The DLT evaluable set included all participants who were evaluable for the DLTs in first cycle and had taken at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-066 0.1 mg/kg | MORAb-066 0.3 mg/kg | MORAb-066 1 mg/kg | MORAb-066 2 mg/kg | MORAb-066 3 mg/kg
Number analyzed (Participants) | 3 | 4 | 5 | 7 | 8
Participants | 0 | 0 | 0 | 1 | 3

3. Secondary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the highest dose level at which no more than one out of six participants experienced DLT. DLT was defined using NCI CTCAE Version 4.03 as any grade 3 or 4 hematemesis, hemoptysis, hematochezia, bright red blood per rectum, epistaxis, gingival bleeding, hemarthrosis, haematuria, uncontrollable menses, or any other bleeding thought to be significant as per assessment of the investigator, regardless of grade.
Time Frame: Cycle 1 (Cycle length=28 days)
Population: as for outcome 2
Measure: Number; unit: mg/kg
Groups:
- MORAb-066: All Participants: Participants received, MORAb-066 0.1 or 0.3 or 1 or 2 or 3 mg/kg, infusion intravenously, on Days 1, 8, 15, and 22, in a 28-day treatment cycle until disease progression, the participant discontinuation due to unacceptable toxicity, withdrawal by participants, or discontinuation by study physician decision.
Arm/Group | MORAb-066: All Participants
Number analyzed (Participants) | 27
mg/kg | 2

4. Secondary Outcome: Cmax: Maximum Observed Serum Concentration for MORAb-066
Time Frame: Cycle 1 Days 1 and 22: 0-168 hours post-dose (Cycle length=28 days)
Population: The pharmacokinetic (PK) analysis set was the group of participants who had sufficient PK data to derive at least one PK parameter. Here, "Number analyzed" signifies participants evaluable at a given time points for this outcome measure.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | MORAb-066 0.1 mg/kg | MORAb-066 0.3 mg/kg | MORAb-066 1 mg/kg | MORAb-066 2 mg/kg | MORAb-066 3 mg/kg
Number analyzed (Participants) | 3 | 4 | 5 | 7 | 8
microgram per milliliter (mcg/mL)
  Cycle 1 Day 1 | 2.09 (0.186) | 5.26 (0.826) | 23.40 (5.697) | 45.65 (12.370) | 68.61 (13.201)
  Cycle 1 Day 22: number analyzed (Participants) | 3 | 2 | 3 | 5 | 2
  Cycle 1 Day 22 | 1.95 (0.731) | 4.33 (0.014) | 21.33 (7.106) | 52.68 (12.544) | 121.50 (30.406)

5. Secondary Outcome: Tmax: Time to Reach Maximum Serum Concentration for MORAb-066
Time Frame: Cycle 1 Days 1 and 22: 0-168 hours post-dose (Cycle length=28 days)
Population: The PK analysis set was the group of participants who had sufficient PK data to derive at least one PK parameter. Here, "Number analyzed" signifies participants evaluable at a given time points for this outcome measure.
Measure: Median (Full Range); unit: hours
Arm/Group | MORAb-066 0.1 mg/kg | MORAb-066 0.3 mg/kg | MORAb-066 1 mg/kg | MORAb-066 2 mg/kg | MORAb-066 3 mg/kg
Number analyzed (Participants) | 3 | 4 | 5 | 7 | 8
hours
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 4 | 5 | 6 | 8
  Cycle 1 Day 1 | 1.28 [1.27 to 3.07] | 1.30 [1.25 to 3.00] | 1.25 [1.02 to 3.00] | 1.80 [1.70 to 3.07] | 1.82 [1.75 to 3.93]
  Cycle 1 Day 22: number analyzed (Participants) | 3 | 2 | 3 | 5 | 2
  Cycle 1 Day 22 | 1.33 [1.25 to 2.00] | 1.25 [1.25 to 1.25] | 1.25 [1.22 to 43.27] | 1.92 [1.37 to 3.52] | 1.77 [1.75 to 1.78]

6. Secondary Outcome: t1/2: Terminal Elimination Phase Half-Life for MORAb-066
Time Frame: Cycle 1 Days 1 and 22: 0-168 hours post-dose (Cycle length=28 days)
Population: The PK analysis set was the group of participants who had sufficient PK data to derive at least one PK parameter. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. Here, "Number analyzed" signifies participants evaluable at a given time points for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MORAb-066 0.1 mg/kg | MORAb-066 0.3 mg/kg | MORAb-066 1 mg/kg | MORAb-066 2 mg/kg | MORAb-066 3 mg/kg
Number analyzed (Participants) | 0 | 2 | 4 | 1 | 1
hours
  Cycle 1 Day 1 |  | 30.8 (10.68) | 52.2 (10.22) | 80.2 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 57.1 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  Cycle 1 Day 22 |  | 24.1 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 44.6 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |  |

7. Secondary Outcome: AUC(0-t): Area Under the Serum Concentration-time Curve From Zero Time to the Last Measurable Point for MORAb-066
Time Frame: Cycle 1 Days 1 and 22: 0-168 hours post-dose (Cycle length=28 days)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours*microgram/milliliter
Arm/Group | MORAb-066 0.1 mg/kg | MORAb-066 0.3 mg/kg | MORAb-066 1 mg/kg | MORAb-066 2 mg/kg | MORAb-066 3 mg/kg
Number analyzed (Participants) | 3 | 4 | 5 | 6 | 8
hours*microgram/milliliter
  Cycle 1 Day 1 | 95.5 (44.92) | 202.3 (41.48) | 1535.6 (589.97) | 2415.5 (1245.84) | 4536.3 (1104.35)
  Cycle 1 Day 22: number analyzed (Participants) | 3 | 2 | 3 | 5 | 2
  Cycle 1 Day 22 | 61.2 (25.09) | 188.5 (51.62) | 1541.3 (1245.66) | 5188.0 (1911.22) | 10420.0 (1244.51)

8. Secondary Outcome: AUC(0-Inf): Area Under the Serum Concentration-time Curve From Zero to Infinity for MORAb-066
Time Frame: Cycle 1 Days 1 and 22: 0-168 hours post-dose (Cycle length=28 days)
Population: The PK analysis set was the group of participants who had sufficient PK data to derive at least one PK parameter. Here,"Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. Here, "Number analyzed" signifies participants evaluable at a given time points for this outcome measure.
Measure: Mean (Standard Deviation); unit: hour*microgram per milliliter
Arm/Group | MORAb-066 0.1 mg/kg | MORAb-066 0.3 mg/kg | MORAb-066 1 mg/kg | MORAb-066 2 mg/kg | MORAb-066 3 mg/kg
Number analyzed (Participants) | 0 | 2 | 4 | 1 | 1
hour*microgram per milliliter
  Cycle 1 Day 1 |  | 249 (4.2) | 1569 (707.9) | 4210 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 5970 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  Cycle 1 Day 22 |  | 227 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 1410 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |  |

9. Secondary Outcome: Vd: Volume of Distribution for MORAb-066
Time Frame: Cycle 1 Days 1 and 22: 0-168 hours post-dose (Cycle length=28 days)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | MORAb-066 0.1 mg/kg | MORAb-066 0.3 mg/kg | MORAb-066 1 mg/kg | MORAb-066 2 mg/kg | MORAb-066 3 mg/kg
Number analyzed (Participants) | 0 | 2 | 4 | 1 | 1
liter
  Cycle 1 Day 1 |  | 5.06 (3.960) | 3.89 (1.029) | 3.88 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 4.01 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  Cycle 1 Day 22 |  | 3.68 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 2.55 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |  |

10. Secondary Outcome: CL: Total Body Clearance for MORAb-066
Time Frame: Cycle 1 Days 1 and 22: 0-168 hours post-dose (Cycle length=28 days)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | MORAb-066 0.1 mg/kg | MORAb-066 0.3 mg/kg | MORAb-066 1 mg/kg | MORAb-066 2 mg/kg | MORAb-066 3 mg/kg
Number analyzed (Participants) | 0 | 2 | 4 | 1 | 1
liter per hour
  Cycle 1 Day 1 |  | 0.1048 (0.05268) | 0.0516 (0.00894) | 0.0362 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 0.0488 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  Cycle 1 Day 22 |  | 0.1060 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 0.0396 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |  |

11. Secondary Outcome: Number of Participants With Best Overall Response (BOR)
Description: BOR based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for target and non-target lesions is complete response (CR) or partial response (PR). CR: disappearance of target and non-target lesions, normalization of tumor marker level, all lymph nodes must be non-pathological in size (less than 10 millimeter [mm] short axis). PR: at least 30 percent (%) decrease in sum of diameters (SOD) of target lesions, taking as reference the baseline SOD persistence of one or more non-target lesions and/or maintenance of tumor marker level above the normal limits. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest SOD. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: Up to approximately 2 years 7 months
Population: The efficacy analysis set was the group of participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-066 0.1 mg/kg | MORAb-066 0.3 mg/kg | MORAb-066 1 mg/kg | MORAb-066 2 mg/kg | MORAb-066 3 mg/kg
Number analyzed (Participants) | 3 | 4 | 5 | 7 | 8
Participants
  Stable Disease | 0 | 0 | 0 | 0 | 1
  Progressive Disease | 3 | 3 | 2 | 3 | 1
  Not Assessed | 0 | 1 | 3 | 4 | 6

12. Secondary Outcome: Number of Participants Positive for Antidrug Antibodies (ADA)
Time Frame: Up to approximately 2 years 7 months
Population: The ADA evaluable population was the participants who received at least one dose of study drug and had at least one post-baseline ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-066 0.1 mg/kg | MORAb-066 0.3 mg/kg | MORAb-066 1 mg/kg | MORAb-066 2 mg/kg | MORAb-066 3 mg/kg
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 4
Participants | 1 | 0 | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: First dose of study drug (Baseline) up to 30 days after last dose of study drug (Up to approximately 2 years 7 months)
Arm/Group | MORAb-066 0.1 mg/kg | MORAb-066 0.3 mg/kg | MORAb-066 1 mg/kg | MORAb-066 2 mg/kg | MORAb-066 3 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/4 | 1/5 | 2/7 | 1/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/4 | 3/5 | 4/7 | 3/8
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 5/5 | 7/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MORAb-066 0.1 mg/kg (N=3) | MORAb-066 0.3 mg/kg (N=4) | MORAb-066 1 mg/kg (N=5) | MORAb-066 2 mg/kg (N=7) | MORAb-066 3 mg/kg (N=8)
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MORAb-066 0.1 mg/kg (N=3) | MORAb-066 0.3 mg/kg (N=4) | MORAb-066 1 mg/kg (N=5) | MORAb-066 2 mg/kg (N=7) | MORAb-066 3 mg/kg (N=8)
Vomiting (Gastrointestinal disorders) | 1 | 2 | 4 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 3 | 2 | 2
Pyrexia (General disorders) | 1 | 0 | 1 | 2 | 2
Chills (General disorders) | 0 | 2 | 1 | 0 | 1
Asthenia (General disorders) | 1 | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 1
Pain (General disorders) | 0 | 0 | 2 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 5 | 6
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 3 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 1 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 3 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0 | 0 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Facial wasting (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes